CLINICAL TRIAL: NCT01104389
Title: A Prospective Investigation of the Use of the Fluorescence Imaging on the da Vinci Surgical System for Intraoperative Near Infrared Imaging of Renal Cortical Tumors
Brief Title: Fluorescence Imaging on the da Vinci Surgical System for Intraoperative Near Infrared Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Song Liu/Clinical Trial Associate, Intuitive Surgical
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ISI-FHU-2010-01
Record Dates: First submitted 2010-04-07; First posted 2010-04-15 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fluorescence imaging — Intraoperatively acquire fluorescence images of renal tumors

SUMMARY:
A Prospective Investigation of the Use of the Fluorescence Imaging on the da Vinci Surgical System for Intraoperative Near Infrared Imaging of Renal Cortical Tumors. To determine the feasibility of the fluorescence imaging on the da Vinci Surgical System in robotic partial nephrectomy procedures and report perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 to 80 years.
* Urine pregnancy test negative for women of childbearing potential prior to surgery
* Subject is able to comply with the study procedures
* A CT or MRI preoperative assessment of renal cortical tumor
* The renal tumor must be stage T1a-b - T2
* Written informed consent.

Exclusion Criteria:

* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests, as total bilirubin >1.5 X normal and/or SGOT >2X normal
* Subject has uremia, serum creatinine >2.0 mg/dl.
* Subject has a previous history of adverse reaction or allergy to ICG, iodine, shellfish or iodine dyes
* Subject in whom the use of x-ray dye or ICG is contraindicated including development of adverse events when previously or presently administered
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Subject is pregnant or lactating
* Subjects actively participating in another drug, biologic and/or device protocol
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
The rate of good or excellent fluorescence images achieved intraoperatively. It will be measured by the correlation of the ultrasound imaging with the fluorescence imaging. | Intraoperatively
  The feasibility of using the fluorescence imaging on the da Vinci Surgical System to detect renal cortical tumors will be measured by the rate of good or excellent images achieved intraoperatively.

SECONDARY OUTCOMES:
Include but not limited to the rate of positive surgical margins, incidence of complications, estimated blood loss and length of stay. | up to 3 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States